CLINICAL TRIAL: NCT06395571
Title: Common Gastrointestinal Symptoms in Healthy Infants Receiving Goat Milk-based Formula or Cow Milk-based Formula: a Double-blind, Randomized Controlled Trial
Brief Title: GI Symptoms in Infants Fed GMF or CMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ausnutria Hyproca B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P19-009
Record Dates: First submitted 2024-04-26; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Gastrointestinal Diseases; Infant Nutrition Disorders
Keywords: goat milk-based infant formula; infant formula; gastrointestinal comfort; infant nutrition
MeSH Terms: conditions — Gastrointestinal Diseases; Infant Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goat milk-based infant formula (Experimental): Experimental group receives goat milk-based formula for 24 weeks
  Interventions: Dietary Supplement: Goat milk-based infant formula
- Cow's milk-based infant formula (Active Comparator): Control group receives cow's milk-based formula for 24 weeks
  Interventions: Dietary Supplement: Cow's milk-based infant formula

INTERVENTIONS:
Dietary Supplement: Goat milk-based infant formula — Goat milk-based infant formula fed at age appropriate quantities for 24 weeks
  Arms: Goat milk-based infant formula
Dietary Supplement: Cow's milk-based infant formula — Cow's milk-based infant formula formula fed at age appropriate quantities for 24 weeks
  Arms: Cow's milk-based infant formula

SUMMARY:
The aim of this study was to assess common gastrointestinal symptoms in healthy Brazilian infants receiving goat milk-based infant formula (GMF) compared to cow's milk-based infant formula (CMF) during a 24 week intervention.

DETAILED DESCRIPTION:
Anecdotal evidence shows that the use of goat milk-based infant formula decreases discomfort of infants with cow's milk related symptoms. In this double-blind, randomized controlled trial, gastrointestinal comfort in infants fed goat milk-based infant formula (GMF) or cow's milk-based infant formula (CMF) was studied.

Fifty-six healthy infants aged 3-12 months were followed for 24 weeks. Stool consistency, regurgitation frequency and crying duration were measured weekly using an adapted version of the Cow's Milk-related Symptom Score (CoMiSS®) where only the items for these scores were used. Blood hemoglobin levels were measured at the start and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* gestational age 37-42 weeks
* 3-12 months old at enrollment
* should have consumed cow's milk-based products during the 48 hours prior to the baseline visit to exclude cow's milk allergic infants

Exclusion Criteria:

* metabolic or chronic disease or congenital malformation, serious concurrent illness that would interfere with study treatment, (i.e. sepsis, pneumonia with respiratory failure, cardiac failure)
* infant's parent(s) or primary caregiver(s) diagnosed with major depression
* infant's weight for length at baseline >|3| z-score indexes according to WHO criteria
* infants enrolled in another interventional clinical research study
* infants diagnosed with cow's milk allergies

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms | 24 weeks, measured weekly
  Stool consistency, regurgitation frequency and crying duration as measured by an adapted Cow's Milk-related Symptom Score®, where a higher score indicates more severe symptoms.

SECONDARY OUTCOMES:
Blood hemoglobin levels | 24 weeks, measured at start and end
  Blood hemoglobin levels before and after intervention
WHO z-score of weight-for-age | 24 weeks, measured monthly
  Weight measured to the nearest 5.0 grams with clothes and diaper removed.
WHO z-score of length-for-age | 24 weeks, measured monthly
  Body length without shoes, measured lying down to the nearest centimeter with a neonatometer.
WHO z-score of head circumference-for-age | 24 weeks, measured monthly
  Head circumference measured with flexible non-stretching tape to the nearest centimeter.
WHO z-score of weight-for-length | 24 weeks, measured monthly
  Weight and length measured as described above combined.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo da Costa Ribeiro, Dr., Principal Investigator — Hospital Professor Edgard Santos, Federal University of Bahia, Salvador, Brazil
Locations (1):
- Daycare center, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maximino P, van Lee L, Meijer-Krommenhoek YN, van der Zee L, da Costa Ribeiro Junior H. Common gastrointestinal symptoms in healthy infants receiving goat milk-based formula or cow's milk-based formula: a double-blind, randomized, controlled trial. BMC Pediatr. 2024 Nov 20;24(1):753. doi: 10.1186/s12887-024-05214-y. PMID 39567910